CLINICAL TRIAL: NCT06154603
Title: Risk Factors for and Survival After Oesophageal, Gastric and Small Intestinal Perforations: a National Observational Registry-based Cohort Study
Brief Title: Upper Gastrointestinal Perforations: a Nationwide Registry-based Study
Status: Not yet recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Rebecka Ahl Hulme, Principle investigator, Region Stockholm
Other Study IDs: K 2023-7938
Record Dates: First submitted 2023-10-12; First posted 2023-12-04 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Acute Abdomen
Keywords: Clinical outcomes; General surgery; Upper gastrointestinal perforation
MeSH Terms: conditions — Abdomen, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Oesophageal perforation: Adult patients (at least 18 years of age) with an oesophageal perforation, treated for it at a Swedish hospital between 2005-2023.
  Interventions: Procedure: Surgical treatment type
- Gastric perforation: Adult patients (at least 18 years of age) with a gastric perforation, treated for it at a Swedish hospital between 2005-2023.
  Interventions: Procedure: Surgical treatment type
- Small intestinal perforation: Adult patients (at least 18 years of age) with a small intestinal perforation, treated for it at a Swedish hospital between 2005-2023.
  Interventions: Procedure: Surgical treatment type

INTERVENTIONS:
Procedure: Surgical treatment type — This observational design will study the clinical outcome for each type of upper gastrointestinal perforation in relation to surgical or non-surgery treatment and in relation to treatment centre.

SUMMARY:
The primary aim of this project is to increase the knowledge about how perforations in the esophagus, stomach and small intestine are treated on a national level. Furthermore, secondary aims include assessment of how different treatment options and type of treating facilities relate to patient survival. This will be done by studying information about all adult patients with an upper GI perforation treated in Sweden during 2005-2023.

ELIGIBILITY:
Inclusion Criteria:

* age of at least 18 years
* perforation in either oesophagus, stomach or small intestine
* treatment carried out in Sweden
* diagnosis set between January 2005 and August 2023

Exclusion Criteria:

* children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with an upper gastrointestinal perforation between 2005-2023 in Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Mortality | One year after diagnosis
  Mortality up to one year after diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Rebecka Ahl Hulme, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No